CLINICAL TRIAL: NCT03950232
Title: An Open-Label Extension Study of Etrasimod in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: An Extension Study for Treatment of Moderately to Severely Active Ulcerative Colitis
Acronym: ELEVATE UC OLE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arena is a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD334-303; C5041012 (Other: Alias Study Number); 2024-515156-21-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06025227 (Available)
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Etrasimod; APD334
MeSH Terms: conditions — Colitis, Ulcerative | interventions — etrasimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Etrasimod 2 mg (Experimental)
  Interventions: Drug: Etrasimod

INTERVENTIONS:
Drug: Etrasimod — Etrasimod 2 mg tablet by mouth, once daily up to approximately 8 years or until marketing authorization is obtained in the participant's country, whichever comes first
  Other Names: APD334

SUMMARY:
The purpose of this open-label extension (OLE) study is to evaluate the safety and efficacy of etrasimod in participants with moderately to severely active ulcerative colitis (UC) who previously received double-blind treatment (either etrasimod 2 mg per day or placebo) during participation in one of the qualified Phase 3 or Phase 2 double-blind, placebo-controlled parent studies including but not limited to: (APD334-301 [NCT03945188] or APD334-302 [NCT03996369] or APD334-210 [NCT04607837]).

ELIGIBILITY:
Inclusion Criteria:

* Must have met the eligibility criteria and have been enrolled in the qualified Phase 2 or 3 parent studies listed below or other qualified region-specific studies and meet the following additional criteria:

  1. Participants previously enrolled in Study APD334-301 (NCT03945188) or APD334-210 (NCT04607837) must have completed the Week 12 visit and have been assessed to have active UC that has not improved or has worsened from baseline or completed the Week 52 visit
  2. Participants previously enrolled in APD334-302 (NCT03996369) must have completed the Week 12 visit

Exclusion Criteria:

* If Investigator considers the participant to be unsuitable for any reason to participate in the Open-Label Extension study
* Experienced an adverse event that led to discontinuation from parent study

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2029-06-19 (Estimated); Study Completion 2029-06-19 (Estimated)

PRIMARY OUTCOMES:
Number and Severity of Safety Measures | Up to approximately 8 years
  Safety as assessed by the evaluation of adverse events

SECONDARY OUTCOMES:
Proportion of Participants Achieving Clinical Remission Assessed by Mayo Component Sub-scores | Week 52 and Week 104
Proportion of Participants Achieving Clinical Remission at Weeks 52 and 104 Among Participants Achieving Clinical Remission at Study Entry | Week 52 and Week 104
Change From Baseline in the Total Mayo Score | Baseline, Week 52, and Week 104
  The total Mayo score is a tool designed to measure disease activity for ulcerative colitis. Scoring ranges from 0 to 12 points and consists of 4 components (endoscopic score, rectal bleeding, stool frequency, and physicians global assessment), each graded 0 to 3 (0 = normal, 1 = mild, 2 = moderate, 3 = severe) with higher score indicating more severe disease.
Change From Baseline in Partial Mayo Score | Baseline, Week 52, Week 104, Week 156, Week 208 and Week 260
  The partial Mayo score is a tool designed to measure disease activity for ulcerative colitis. Scoring ranges from 0 to 9 points and consists of 3 non-invasive components (rectal bleeding, stool frequency, and physicians global assessment), each graded 0 to 3 (0 = normal, 1 = mild, 2 = moderate, 3 = severe) with higher score indicating more severe disease.
Proportion of Participants Achieving Endoscopic Improvement Assessed by Mayo Component Sub-scores | Week 52 and Week 104
Proportion of Participants Achieving Clinical Response Assessed by Mayo Component Sub-scores | Week 52 and Week 104

OTHER OUTCOMES:
Percentage of Participants With Histologic Improvement Assessed by the Geboes, Robarts, and Nancy Histopathology Scores | Week 52 and Week 104
Percentage of Participants With Histologic Remission Assessed by the Geboes, Robarts, and Nancy Histopathology Scores | Week 52 and Week 104
Time to Loss of Response Assessed by Mayo Component Sub-scores | Up to Week 260
Proportion of Participants Achieving Improvement in Extraintestinal Manifestations (EIMs) in Participants With EIMs at Baseline | Baseline, Week 12, Week 52, Week 104, Week 156, Week 208, and Week 260

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (461):
- United States (124):
  - Center for Digestive Health (Colonoscopy Location), Dothan, Alabama
  - Pulmonary Associates (Secondary PFT Location), Dothan, Alabama
  - Gut P.C., dba Digestive Health Specialists of the Southeast (IP Address), Dothan, Alabama
  - Inland Pulmonary Specialists [PFT Only], Lake Elsinore, California
  - A V Pediatrics,Allergy and Family Medicine, Lancaster, California
  - Advanced Endoscopy and Pain Center(Colonoscopy), Lancaster, California
  - Antelope Valley Eye Care(Ophthalmologist), Lancaster, California
  - Jatinder S.Pruthi,MD FACG CPI, Lancaster, California
  - Om Research LLC, Lancaster, California
  - Renaissance Imaging Center(Chest X-Ray only), Lancaster, California
  - United Surgery Center Murrieta [Endoscopy Only], Murrieta, California
  - United Medical Doctors, Murrieta, California
  - Advanced Imaging (Chest X-Ray), Palmdale, California
  - California Eye Professionals [OCT Only], Temecula, California
  - United Surgery Center Temecula [Endoscopy Only], Temecula, California
  - Front Range Endoscopy Center, Colorado Springs, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Bay Area Chest Physicians, P.A.,-(Pulmonary Function Test), Clearwater, Florida
  - West Coast Endoscopy Center (Endoscopy Procedures), Clearwater, Florida
  - Northwood Vision-Optical Coherence Tomography-(OCT), Clearwater, Florida
  - Safety Harbor Surgery (Endoscopy Facility), Clearwater, Florida
  - Gastro Florida (Regulatory & Administrative Duties), Clearwater, Florida
  - Gastro Florida-(Regulatory & Administrative Duties), Clearwater, Florida
  - Dr Lee Shettle, Largo, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - Tampa Bay Regional Surgery Center, Largo, Florida
  - NSB Research, New Smyrna Beach, Florida
  - Tampa Bay Endoscopy Center (ENDO Only), Tampa, Florida
  - Tampa Bay Endoscopy Center, Tampa, Florida
  - Lab - Processing / Storage, Tampa, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - Pulmonary and Sleep of Tampa Bay (PFT Only), Tampa, Florida
  - GCP Clinical Research,LLC, Tampa, Florida
  - LoCicero Medical Group (PFT Procedure Only), Tampa, Florida
  - Lyracore Health Alliance (PFT Procedure only), Tampa, Florida
  - Newsome Eye Specialist (OCT Procedures Only), Tampa, Florida
  - USF Health Morsani Center For Advanced Healthcare, Tampa, Florida
  - Guardian Angel Research Center, INC, Tampa, Florida
  - Perez Eye Center (OCT only), Tampa, Florida
  - Florida Medical Clinic, LLC (Endoscopy), Zephyrhills, Florida
  - Florida Medical Clinic, LLC (OCT), Zephyrhills, Florida
  - Florida Medical Clinic, LLC (PFT), Zephyrhills, Florida
  - Florida Medical Clinic, LLC, Zephyrhills, Florida
  - Emory Pulmonary Function Tedt Lab, Atlanta, Georgia
  - Emory Pulmonary Group (PFT only), Atlanta, Georgia
  - Atlanta Gastroenterology Associates (Endoscopy Location), Atlanta, Georgia
  - Atlanta Gastroenterology Associates (Screening and Recruitment), Atlanta, Georgia
  - Atlanta Gastroenterology Associates(IP only), Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Emory Saint Joseph Pulmonary Function Test Lab, Atlanta, Georgia
  - Thomas Eye Group (OCT only), Sandy Springs, Georgia
  - Illinois Gastroenterology Group dba GI Alliance (Patients seen; IP Delivered), Gurnee, Illinois
  - Medical Eye Services LTD (Ophthalmoscopy with OCT), Gurnee, Illinois
  - North Shore Endoscopy Center (Endoscopy), Lake Bluff, Illinois
  - Libertyville Imaging Center (Diagnostic Imaging), Libertyville, Illinois
  - Eye Medical Center (OCT location), Baton Rouge, Louisiana
  - Baton Rouge LA Endoscopy, Baton Rouge, Louisiana
  - Chevy Chase Pulmonary Associate (PFT Only), Chevy Chase, Maryland
  - Retina Group Of Washington (OCT Only), Chevy Chase, Maryland
  - Barnes-Jewish West County Hospital (Additional Endoscopy Location), Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Durango Surgical Center, Las Vegas, Nevada
  - Abrams Eye Institute (OCT), Las Vegas, Nevada
  - Lung Center of Nevada, Las Vegas, Nevada
  - Duke Medical Plaza North Duke Street, Durham, North Carolina
  - Duke Eye Center (OCT only), Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Investigational Drug Services (Pharmacy), Durham, North Carolina
  - Brier Creek Medical Pavilion, Raleigh, North Carolina
  - Geauga Sleep Center (PFT Only), Chardon, Ohio
  - UC Health Hoxworth (OCT only), Cincinnati, Ohio
  - UC Health Physicians Office, Cincinnati, Ohio
  - University of Cincinnati Medical Center (PFT and Endoscopy location), Cincinnati, Ohio
  - University of Cincinnati Medical Center Investigational Pharmacy, Cincinnati, Ohio
  - UC Health (Pulmonary Function Testing), Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Ophthalmic Physicians Incorporated (OCT Only), Mentor, Ohio
  - The Endoscopy Center of Lake County, Mentor, Ohio
  - Vitreo Retinal Consultants (OCT only), Mentor, Ohio
  - Lake Pulmonary Associates (PFT only), Willoughby Hills, Ohio
  - Retina Specialist of Ohio (OCT only), Willoughby Hills, Ohio
  - Digestive Disease Specialists, Inc. Endoscopy Lab, Oklahoma City, Oklahoma
  - Pulmonary Physicians of Oklahoma, Oklahoma City, Oklahoma
  - Retina Center of Oklahoma, Oklahoma City, Oklahoma
  - Susquehanna Research Group, Camp Hill, Pennsylvania
  - West Shore Endoscopy Center, Camp Hill, Pennsylvania
  - Farrell Ophthalmology (OCT only), Harrisburg, Pennsylvania
  - Susquehanna Research Group, LLC, Harrisburg, Pennsylvania
  - Harrisburg Eye Associates (OCT only), Harrisburg, Pennsylvania
  - Medical Arts Allergy,PC (PFT Only), Harrisburg, Pennsylvania
  - Pulmonary and Critical Care Medicine Associates (PFT only), Lemoyne, Pennsylvania
  - Cross Timbers Surgery Center(Proctosigmoidoscopy), Arlington, Texas
  - Envision Imaging(Chest X-Ray), Arlington, Texas
  - Texas Clinical Research Institute, Arlington, Texas
  - Texas Pulmonary and Critical Care Associates(Pulmonary Function Test), Arlington, Texas
  - Texas Retina Associates(Ophthalmoscopy), Arlington, Texas
  - Inquest Clinical Research, Baytown, Texas
  - Texas Retina Associates (OCT Location), Grapevine, Texas
  - Plaza Medical Center, Houston, Texas
  - East Houston Physicians Group, Houston, Texas
  - Baylor College of Medicine- Baylor Medical Center, Houston, Texas
  - Cross Eye Center (Optical Coherence Tomography), Houston, Texas
  - Lonestar Endoscopy(Endoscopy Location), Keller, Texas
  - Christus Santa Rosa Physicians Ambulatory Surgery Center New Braunfels (Endoscopy), New Braunfels, Texas
  - Tyrus Schroeder (PFT), New Braunfels, Texas
  - Central Texas Eye Center (OCT), San Marcos, Texas
  - Christus Santa Rosa Physicians Ambulatory Surgery Center San Marcos (Endoscopy), San Marcos, Texas
  - Envision Imaging (Chest X-ray location), Southlake, Texas
  - Lonestar Endoscopy (Endoscopy Location), Southlake, Texas
  - Christus Trinity Mother Frances Endosopy Center ( endoscopies only), Tyler, Texas
  - Heaton Eye Associates (OCT only), Tyler, Texas
  - UT Health East Texas Physicians (pulmonary functions only), Tyler, Texas
  - Gastro Health & Nutrition, Victoria, Texas
  - Harman Eye Center (OCT only), Forest, Virginia
  - Lynchburg Pulmonary Associates, Inc. (PFT only), Lynchburg, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Swedish Endoscopy Center - Issaquah, Issaquah, Washington
  - Pacific Northwest Retina, Seattle, Washington
  - Richard Bensinger, MD, Seattle, Washington
  - Swedish Gastroenterology, Seattle, Washington
  - Swedish Medical Center First Hill Endoscopy Center, Seattle, Washington
  - Swedish Medical Center First Hill, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Centro de lnvestigation C.I .C.E. 9 de Julio, San Miguel de Tucumán, Tucumán Province, Argentina
- Australia (11):
  - Liverpool Hospital, Liverpool, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Coral Sea Clinical Research Institute Pty.Ltd, Mackay, Queensland
  - Dr Shiran DeSilva Respiratory Clinic, Mackay, Queensland
  - Mackay Discount Drug Store, Mackay, Queensland
  - Mater Misericordiae Hospital, Mackay, Queensland
  - Queensland X-Ray, Mackay, Queensland
  - Vision Eye Institute Mackay, Mackay, Queensland
  - Coastal Digestive Helath Pty. Ltd, Maroochydore, Queensland
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Department of Internal Medicine III, Clinical Division of Gastroenterology and Hepatology, Vienna, Austria
- Belarus (9):
  - Foreign Medical and Pharmaceutical Unitary Enterprise "Medical Center" Novoe Zrenie", Grodno
  - Health Care Institution "City Clinical Hospital #4 Grodno", Grodno
  - Healthcare Institution "Grodno University Hospital", Grodno
  - Institution "Gomel Regional Specialized Clinical Hospital", Homyel
  - Institution "Gomel Regional Clinical Hospital, Homyel
  - Health care Institution "10th City Clinical Hospital", Minsk
  - Educational Establishment "Vitebsk State Medical University", Vitebsk
  - Health Care Institution "Vitebsk Regional Clinical Hospital", Vitebsk
  - Healthcare Institution: Vitebsk Regional Clinical Specialized Center, Vitebsk
- Belgium (3):
  - Hospital AZ Sint-Lucas, Ghent
  - AZ Delta campus Brugsesteenweg, Roeselare
  - AZ Delta, Roeselare
- Bulgaria (10):
  - "UMHAT "Kanev"" AD, Ruse, Rousse
  - Diagnostic-Consultative Center I - Sliven, EOOD, Sliven
  - Acibadem City Clinic Tokuda Hospital EAD, Sofia
  - Acibadem City clinic University Hospital EOOD, Sofia
  - "DCC Alexandrovska", EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski" EAD', Sofia
  - UMHAT "Tsaritsa Yoanna - ISUL" EAD, Sofia
  - "University multiprofile hospital for active treatment and emergency medicine N.I. Pirogov"EAD, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - Medical Centre MEDICA Plus OOD, Veliko Tarnovo
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Clinical Research Chile, Valdivia, Los Ríos Region, Chile
- Croatia (2):
  - General Hospital Zadar, Zadar
  - University Hospital Center Zagreb, Zagreb
- Czechia (14):
  - Gastroenterologicka ambulance, Nemocnice Boskovice, Boskovice
  - Fakultni nemocnice u svate Anny v Brne, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - GASTRO JeKa, s.r.o., Klatovy
  - Endoskopicke pracoviste, Interni oddeleni, Olomouc
  - Ocni ordinace Olomouc (OCT/ophtalmoscopy), Olomouc
  - PreventaMed s.r.o., Olomouc
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Axon Clinical, s.r.o., Prague
  - Nemocnice Na Bulovce, Prague
  - ISCARE a.s., Prague
  - Gastroenterologie, MUDr. Michal Konecny, Ph.D., s.r.o., Přerov
  - Nemocnice Slany, Slaný
  - GASTRO-NELL s.r.o., MUDr. Vladimir Vaculin, Vsetín
- Denmark (2):
  - Aalborg University Hospital, department of medical gastroenterology,, Aalborg
  - Herlev Hospital, Stomach, -Bowel and Liver disease, Clinic 1, Herlev
- Estonia (6):
  - Innomedica OÜ, Tallinn, Harju
  - OCT: Eye Clinic Dr. Krista Turman, Tallinn
  - DLCO: East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Endoscopy: North Estonia Medical Centre Foundation, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
- France (15):
  - CHU Amiens Picardie, Amiens
  - Endoscopy: CHU Amiens-Picardie, Amiens
  - Pulmonary examination: CHU Amiens-Picardie, Amiens
  - Tomography: CHU Amiens-Picardie, Amiens
  - CHU Grenoble Alpes -Hopital Michallon, Grenoble
  - Endoscopy: CHU Grenoble Alpes- Hopital Michallon, Grenoble
  - Pulmonary examination: CHU Grenoble Alpes - Hopital Michallon, Grenoble
  - Tomography: CHU Grenoble Alpes - Hopital Michallon, Grenoble
  - CHU Montpellier Hopital Saint-Eloi, Montpellier
  - Endoscopy: Hopital Saint-Eloi, Montpellier
  - Pulmonary examination: Hopital Arnaud de Villeneuve, Montpellier
  - CHU Hotel Dieu, Nantes
  - CHU de Nice - Hopital de l'Archet 2, Nice
  - CHU de Toulouse-Hopital Rangueil, Toulouse
  - Tomography: CHU RANGUEIL, Toulouse
- Georgia (9):
  - LLC Todua Clinic, Tbilisi
  - Israeli-Georgian Medical Research Clinic Helsicore, LTD, Tbilisi
  - LLC Vivamedi, Tbilisi
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Institute of Clinical Cardiology, Tbilisi
  - Medical Center CITO LTD, Tbilisi
  - LTD Academician Nikoloz Kipshidze Central University Clinic, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center, LTD, Tbilisi
- Germany (7):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte Medizinische Klinik m. S. Hepatologie, Berlin
  - Dr. med Zacharias A. R.Sherif, Berlin
  - Krankenhaus Waldfriede e.V.,, Berlin
  - Schwerpunktpraxis Bonn, Bonn-Duisdorf
  - Johanna-Etienne-Krankenhaus, Neuss
  - OCT address: AOZNeuss Dr. Kersten, Neuss
  - Praxis Dr. Jorgensen, Remscheid
- Hungary (14):
  - Ophthalmology tests:Bekes Megyei Kozponti Korhaz, Pady Kalman Tagkorhaz, Szemeszeti Osztaly, Gyula, Bekes County
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár, Fejér
  - Clinfan Szolgaltato Kft., Szekszárd, Tolna County
  - Ophthalmology tests: Tolna Megyei Balassa Janos Korhaz, Szekszárd, Tolna County
  - Endoscopy: Magyar Imre Korhaz, Ajka, Veszprém megye
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred, Veszprém megye
  - Pulmonary function tests, endoscopy: Deak Jeno Korhaz, Tapolca, Veszprém megye
  - Békés Vármegyei Központi Kórház Dr. Réthy Pál Tagkórház, Békéscsaba
  - Pulmonary function tests: Vasutegeszsegugyi Nonprofit Kozhasznu Kft., Budapest
  - Ophthalmology tests: Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Gyöngyösi Bugát Pál Kórház, Gyöngyös
  - Ophthalmology tests: RETINASZERVIZ Kft., Veszprém
- India (8):
  - Sids Hospital & Research Centre, Surat, Gujarat
  - Surat Institute of Digestive Sciences, Surat, Gujarat
  - Fortis Memorial Research Institute, Gurgaon, Haryana
  - Midas Multispeciality Hospital Pvt. Ltd, Nagpur, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - S.R.Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Post Graduate Department Of Medicine, Kanpur, Uttar Pradesh
  - Government Medical College & Super Speciality Hospital, Nagpur
- Israel (7):
  - Bnai Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Galilee Medical Center, Naharya
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Italy (13):
  - I.R.C.C.S "Saverio De Bellis", Gastroenterologia II, Castellana Grotte, BARI
  - Spedali Civili di Brescia, U.O. Gastroenterologia, Brescia, Lombardy
  - IRCCS Ospedale San Raffaele, Oculistica, Milan, Lombardy
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese, Milano
  - ASST Rhodense - U.O.C. di Gastroenterologia ed Endoscopia Digestiva, Rho, Milan
  - A.O.U. Policlinico di Modena, Modena, Reggio Emilia
  - Azienda Ospedaliero Universitaria Careggi, U.O. Gastroenterologia 2 (St.19), Florence, Tuscany
  - Ospedale Sacro Cuore Don Calabria, Negrar(vr), VR
  - Azienda Ospedalieria Ospedale Cannizzaro, Catania
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro
  - IRCCS Ospedale San Raffaele UO di Gastroenterologia e Endoscopia Digestiva, Milan
  - U.O.C. Gastroenterologia ed Endoscopia Digestiva, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS -CEMAD -UOC di Medicina lnterna e Gastro, Roma
- Japan (57):
  - Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Kojunkai Daido Hospital, Nagoya, Aixhi-ken
  - Tsujinaka Hospital Kashiwanoha, Kashiwa-shi, Chiba
  - Ishii Eye Clinic, Nagareyama-shi, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Fukuoka Tokushukai Hospital, Kasuga, Fukuoka
  - Takimoto Eye Clinic(OCT), Kasuga-shi, Fukuoka
  - Japan Community Health Care Organization Kyushu Hospital, Kitakyushu, Fukuoka
  - Koyanose Eye Clinic, Kitakyushu-shi, Fukuoka
  - Our Lady of the Snow St. Mary's Hospital, Kurume, Fukuoka
  - Fukuoka Shinmizumaki Hospital, Onga-gun, Fukuoka
  - Gifu University Hospital, Gifu, Gifu
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ota-shi, Gunma
  - National Hospital Organization Fukuyama Medical Center, Fukuyama, Hiroshima
  - Nakayama EYE Clinic, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Asahikawa City Hospital, Asahikawa-shi, Hokkaido
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - NHO Mito Medical Center, Higashiibaraki-gun, Ibaraki
  - Matsumoto Eye Clinic, Toride-shi, Ibaraki
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Iwate Medical University Uchimaru Medical Center, Morioka, Iwate
  - Kagawa Prefectural Central Hospital, Takainatsu-shi, Kagawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - JA- Kagoshima Koseiren Hospital (PET/DLCO), Kagoshima, Kagoshima-ken
  - Jiaikai Idzuro Imamura Hospital, Kagoshima, Kagoshima-ken
  - Sameshima Eye Clinic (OCT), Kagoshima, Kagoshima-ken
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Social Welfare Organization Imperial Gift Foundation,Inc.Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Hinaga Nishi Ophthalmology Clinic, Yokkaichi- Shi, Mie-ken
  - Mie Prefectural General Medical Center, Yokkaichi-shi, Mie-ken
  - JOHAS Tohoku Rosai Hospital, Sendai, Miyagi
  - Sendai City Hospital, Sendai, Miyagi
  - Nagaoka Red Cross Hospital, Nagaoka-shi, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Japan Community Health care Organization Osaka Hospital, Osaka, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Matsuda Hospital, Hamamatsu, Shizuoka
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka
  - St. Luke's International Hospital, Chuo-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Showa General Hospital, Kodaira-shi, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Wakayama Medical University Hospital, Wakayama, Wakayama
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Fukushima Medical University Hospital, Fukushima
  - Kansai Medical University Hospital, Hirakata
  - NHO Osaka National Hospital, Osaka
  - Saga University Hospital, Saga
- P. Stradins Clinical University Hospital, Gastroenterology, Hepatology and Nutrition Therapy Center, Riga, Latvia
- American University of Beirut Medical Center, Beirut, Lebanon
- Lithuania (5):
  - Consultancy Polyclinic of Republican Panevezys Hospital, Panevezys
  - Republican Panevezys Hospital, Panevezys
  - UAB "Northway", Medical and Surgical Centre, Vilnius
  - UAB "Inlita", Santaros Clinical Trials Centre, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (8):
  - Invesclinic MX, Irapuato, Guanajuato
  - Centro de lnvestigacion Medico Biologica y Terapia Avanzada S.C., Guadalajara, Jalisco
  - Servicios Medicos y de lnvestigacion Clinica Inspirepharma S. de R.L. de C.V., Monterrey, Nuevo León
  - Scientia, Investigacion Clinica S.C., Chihuahua City
  - Scientia Investigación Clínica S.C, Chihuahua City
  - Invesclinic MX, Irapuato
  - FAICIC S. de R.L. de C.V., Veracruz
  - Servicios Medicos y de lnvestigacion Clinica Inspirepharma S. de R.L. de C.V., Veracruz
- Moldova (4):
  - IMSP Institutul de Ftiziopneumologie "Chiril Draganiuc", Chisinau
  - IMSP Spitalul Clinic Republican "Timofei Mosneaga", Chisinau
  - ISMP Spitalul Clinic Republican "Timofei Mosneaga", RTL SM, Chisinau
  - Spitalul Polivalent Novamed, Chisinau
- Poland (22):
  - NSZOZ Termedica - Centrum Badan Klinicznych, Poznan, Greater Poland Voivodeship
  - Centrum Dentystyczno-Lekarskie PROMEDICA Joanna Markiewicz, Będzin
  - Centrum Medycyny Oddechowej, Mroz Spolka Jawna (PFT, DLCO), Bialystok
  - Gastromed Kralisz, Romatowski, Stachurska sp.j., Bialystok
  - LSSP Eskulap (OCT, Ophthalmoscopy), Bialystok
  - Dobry Wzrok (OCT), Gdansk
  - Poradnia Pulmonologiczna, Gdynia
  - Karkonoskie Centrum Badan Klinicznych - Lexmedica Spolka z ograniczona odpowiedzialnoscia, Jelenia Góra
  - PROMED Centrum Medyczne (OCT, ophthalmoscopy), Jelenia Góra
  - IP Clinic Sp. z o.o., Lodz
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Allmedica Badania Kliniczne Sp. z o.o. Sp. k., Nowy Targ
  - MEDICOME Sp. z o.o., Oświęcim
  - Centrum Medyczne MEDYK, Rzeszów
  - ENDOSKOPIA Sp. z o.o., Sopot
  - DC-MED Sp. z o.o., Swidnica
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych Administracji, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnia we Wroclawiu, Wroclaw
  - Amicare Sp. z o.o. Sp.k., Lodz, Łódź Voivodeship
- Portugal (4):
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE, Vila Nova de Gaia, Porto District
  - Centro Hospitalar e Universitario de Coimbra, EPE, Coimbra
  - Hospital Senhora da Oliveira Guimaraes, E.P.E, Guimarães
  - Centro Hospitalar Universitario de Sao Joao, E.P.E, Porto
- Romania (8):
  - SC Pelican lmpex SRL, Oradea, Bihor County
  - Oculens Med S.R.L., Cluj-Napoca, Cluj
  - Monza Oncology Hospital. Gastroenterology Department, Bucharest, District 1
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca, JUD. CLUJ
  - S.C. Euroclinic Hospital S.A., Bucharest, Sector 1
  - S.C. Euroclinic Hospital S.A., Bucharest
  - Spitalul de Oncologie Monza, Bucharest
  - Spitalul Clinic de Pneumoftiziologie Leon Daniello Cluj-Napoca, Cluj-Napoca
- Russia (27):
  - LLC "Multidisciplinary Medical Clinic "Anturium", Barnaul, Altayskiy Kray
  - LLC Medical Company "Hepatologist", Samara, Samara Oblast
  - LLC "Polyclinic of ultrasonography 4D", Pyatigorsk, Stavropol Kray
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - Professional Education" of MoH of RF, Irkutsk
  - LLC "Alliance Biomedical -Ural Group", Izhevsk
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - State Budgetary Healthcare Instit. of Nizhniy Novgorod region, Nizhny Novgorod
  - LLC "SibNovoMed", Novosibirsk
  - LLC "Novosibirsk GastroCenter", Novosibirsk
  - State Budgetary Healthcare Institution of Novosibirsk region "City clinical hospital # 12", Novosibirsk
  - Medical center "AVITSENNA", Novosibirsk
  - Clinicodiagnostic center "Ultramcd", Omsk
  - State Budgetary Healthcare Institution "Penza Region Clinical Hospital n.a. N.N. Burdenko", Penza
  - Federal State Budgetary Ed. Inst. of Higher Education "North-Western Medical University n.a. I.I., Saint Petersburg
  - FSBEI of Higher Education "North-Western State Medical University n.a. I.I. Mechnikov" of MoH RF, Saint Petersburg
  - Spb SBIH "City Mariinskaya Hospital", Saint Petersburg
  - LLC "Medi com" (SM-Clinic), Saint Petersburg
  - FSBEI of Higher Education "First Saint Petersburg State Medical University n.a. I.P. Pavlov", Saint Petersburg
  - LLC "Gastroenterological centre Expert", Saint Petersburg
  - St.Petersburg State Budgetary Healthcare Institution "City Hospital #40 of Kurortnyi region", Saint Petersburg
  - Private Educational Institution of Higher Education "Medical University "Reaviz", Multifield Clinic, Samara
  - LLC Medical company "Hepatologist", Samara
  - Autonomous Noncommercial Medical Organizations "Stavropol Regional Clinical Diagnostic Centre'', Stavropol
  - Autonomous Noncommercial Medical Organizations " Stavropol Regional Clinical Diagnostic Centre '', Stavropol
  - City Polyclinic #9, Stavropol
  - State Healthcare Institution of Yaroslavl Region "Clinical Hospital No 2", Yaroslavl
- Serbia (3):
  - Clinical Center " Dr Dragisa Misovic-Dedinje", Belgrade
  - Clinical Center Zvezdara, Belgrade
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
- Slovakia (15):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, II. Interna klinika SZU, Banská Bystrica
  - DEJA. s.r.o .. Oftalmologicka ambulancia, Bardejov
  - ALIAN, s.r.o., Bardejov
  - 3F, s.r.o., Oftalmologicka ambulancia, Košice
  - OCULOSANUS, s.r.o., Oftalmologicka ambulancia, Levice
  - MUDr. Michal Popovec, s.r.o., Oftalmologicka ambulancia, Lipany
  - KM Management, spol. s r.o .. Gastroenterologicke a hepatologicke centrum, Nitra
  - Fakultna nemocnica Nitra, Oftalmologicka ambulancia, Nitra
  - Fakultna nemocnica Nitra, Pneumologicka ambulancia, Nitra
  - Fakultna nemocnica Nitra, Nitra
  - GASTRO I., s.r.o. Gastroenterologicka ambulancia, Prešov
  - PULMO, s.r.o., Plucna ambulancia, Prešov
  - Accout Center, s.r.o., Gastroenterologicka ambulancia, Šahy
  - COR, s.r.o., Pneumologicko-ftizeologicka ambulancia, Šahy
  - PULMOX spol. s r.o., Pneumologicko-ftizeologicka ambulancia, Vranov nad Topľou
- South Africa (4):
  - Johese Clinical Research:Unitas, Centurion, Gauteng
  - Unitas Hospital, Centurion, Gauteng
  - Dr John Philip Wright, Cape Town, Western Cape
  - Dr Fritz Potgieter, Midstream Medi Clinic, Centurion
- South Korea (12):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Endoscopy Facility in The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - OCT Facility in The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - PFT Facility in The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - OCT Facility in Dong-A University Hospital, Busan
  - Endoscopy Facility in Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - OCT Facility in Kyungpook National University Chilgok Hospital, Daegu
  - PFT Facility in Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
- Spain (2):
  - HOSPITAL GENERAL UNIVERSITARIO de Alicante, Alicante, Valencia
  - Hospital Universitario la Paz, Madrid
- Thailand (3):
  - Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok
  - Chulalongkorn University, King Chulalongkorn Memorial Hospital, Pathumwan, Bangkok
  - Chulalongkorn University, King Chulalongkorn Memorial Hospital, Bangkok
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Saglik Bilimleri Universitesi Antalya Egitim ve Arastirma Hastanesi, Antalya
  - Uludag University Medical Faculty, Bursa
  - Kocaeli University Medical Faculty, Kocaeli
- Ukraine (19):
  - Communal Institution I.I. Mechnykov Dnipropetrovsk Regional Clinical Hospital, Department of, Dnipro
  - Communal Non-commercial Enterprise Regional Clinical Hospital of lvano-Frankivsk Regional Council,, Ivano-Frankivsk
  - Municipal Health Care "Kharkiv City Hospital Ambulance and Emergency Medical care named alter prof., Kharkiv
  - Llc "Ldts-Skaymed", Kharkiv
  - LLC "EyeQClinic", Kharkiv
  - Communal Noncommercial Enterprise Prof. O.O.Shalimov City Clinical Hospital #2 of Kharkiv City, Kharkiv
  - Llc Medical Center Oftalmika, Kharkiv
  - Communal Noncommercial Enterprise City Clinical Hospital # 13 of Kharkiv City Council,, Kharkiv
  - Communal Noncommercial Enterprise Ye.Ye. Karabelesh Kherson City, Kherson
  - LLC "Diagnostic center", Kherson
  - Kyiv City Clinical Hosptial #1, Department of Therappy #2, Kyiv
  - Communal Noncommercial Enterprise Lviv Clinical Emergency Hospital, 1st Department of Therapy, Lviv
  - Communal Institution Odesa Regional Clinical Hospital, Regional Center of Gastroenterology,, Odesa
  - LLC GLB Clinik, Odesa
  - Andrii Novak Transcarpathian Regional Clinical Hospital, Department of Gastroenterology, Uzhhorod
  - Medical Clinical Investigational Center of Med Center LLC Health Clinic, Unit of Gastroenterology,, Vinnytsia
  - Communal Nonprofit Enterprise M.I.Pyrogov Vinnytsia Regional Clinical Hospital of Vinnytsia Regional, Vinnytsia
  - Scientific and Research Institute of Invalid Rehabilitation (Educational and Scientific Treatment, Vinnytsia
  - Llc "Optimal M", Vinnytsia
- United Kingdom (3):
  - Yeovil District Hospital NHS Foundation Trust, Yeovil, Somerset
  - Barts Health NHS Trust - Whipps Cross University Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Vermeire S, Rubin DT, Peyrin-Biroulet L, Dubinsky MC, Regueiro M, Irving PM, Goetsch M, Lazin K, Gu G, Wu J, Modesto I, McDonnell A, Guo X, Green J, Dalam AB, Yarur AJ. Cardiovascular events observed among patients in the etrasimod clinical programme: an integrated safety analysis of patients with moderately to severely active ulcerative colitis. BMJ Open Gastroenterol. 2025 Jan 8;12(1):e001516. doi: 10.1136/bmjgast-2024-001516. PMID 39778975
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=APD334-303